CLINICAL TRIAL: NCT01649375
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study of Subcutaneous Secukinumab in Prefilled Syringes to Demonstrate Efficacy at 16 Weeks and to Assess Long-term Efficacy, Safety and Tolerability up to 5 Years in Patients With Active Ankylosing Spondylitis
Brief Title: 16 Week Efficacy and 5 Year Long Term Efficacy, Safety and Tolerability of Secukinumab in Patients With Active Ankylosing Spondylitis
Acronym: MEASURE2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2310; 2012-000046-35 (EudraCT Number)
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Anklyosing Spondylitis
Keywords: Ankylosing spondylitis; AS; Chronic inflammatory disease; Inflammatory back pain; Secukinumab; Prefilled syringe; PFS; Subcutaneous injection; AIN457; AIN457F; AIN457F2310; adult
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Secukinumab 75 mg (Experimental): Secukinumab 75 mg subcutaneous injection once weekly at baseline, Weeks 1, 2, 3 and 4, followed by dosing every 4 weeks.
  Interventions: Drug: Secukinumab (75 mg)
- Secukinumab 150 mg (Experimental): Secukinumab 150 mg subcutaneous injection once weekly at baseline, Weeks 1, 2, 3 and 4, followed by dosing every 4 weeks
  Interventions: Drug: Secukinumab (150 mg)
- Placebo (Placebo Comparator): Placebo subcutaneous injection once weekly at baseline, Weeks 1, 2, 3 and 4, followed by dosing every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab (75 mg) — Secukinumab 75 mg s.c.
  Other Names: AIN457 75 mg
  Arms: Secukinumab 75 mg
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Secukinumab (150 mg) — Secukinumab 150 mg s.c.
  Other Names: AIN457 150 mg
  Arms: Secukinumab 150 mg

SUMMARY:
This study assessed the efficacy and safety of secukinumab in patients with active ankylosing spondylitis who were tolerant to or had an inadequate response to NSAIDs, DMARDs and / or TNFα inhibitor

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female patients
* Diagnosis of moderate to severe AS with prior documented radiologic evidence (x-ray) fulfilling the Modified New York criteria for AS (1984)
* Patients should have been on NSAIDs with an inadequate response
* Patients who were regularly taking NSAIDs as part of their AS therapy are required to be on a stable dose
* Patients who had been on an anti-TNFα agent (not more than one) must have experienced an inadequate response

Exclusion Criteria:

* Chest X-ray (or MRI) with evidence of ongoing infectious or malignant process
* Patients with total ankylosis of the spine
* Patients previously treated with any biological immunomodulating agents except for those targeting TNFα
* Previous treatment with any cell-depleting therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2012-10-18 (Actual); Primary Completion 2014-08-04 (Actual); Study Completion 2018-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (49):
- United States (9):
  - Novartis Investigative Site, Mesa, Arizona
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Tupelo, Mississippi
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Mesquite, Texas
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Canada (4):
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Pointe-Claire, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Czechia (4):
  - Novartis Investigative Site, Bruntál, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Uherské Hradiště
- Finland (5):
  - Novartis Investigative Site, HUS, Finland
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Hyvinkää
  - Novartis Investigative Site, Jyväskylä
  - Novartis Investigative Site, Seinäjoki
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Würzburg
- Italy (3):
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Verona, VR
- Netherlands (2):
  - Novartis Investigative Site, Utrecht, The Netherlands
  - Novartis Investigative Site, Amsterdam
- Russia (6):
  - Novartis Investigative Site, Korolyov
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Singapore, Singapore
- Spain (3):
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Madrid
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Fribourg
  - Novartis Investigative Site, Zurich
- United Kingdom (4):
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Torquay

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Marzo-Ortega H, Sieper J, Kivitz AJ, Blanco R, Cohen M, Pavelka K, Delicha EM, Stefanska A, Richards HB, Rohrer S. 5-year efficacy and safety of secukinumab in patients with ankylosing spondylitis: end-of-study results from the phase 3 MEASURE 2 trial. Lancet Rheumatol. 2020 Jun;2(6):e339-e346. doi: 10.1016/S2665-9913(20)30066-7. PMID 38273597
- [Derived] Dougados M, Kiltz U, Kivitz A, Pavelka K, Rohrer S, McCreddin S, Quebe-Fehling E, Porter B, Talloczy Z. Nonsteroidal anti-inflammatory drug-sparing effect of secukinumab in patients with radiographic axial spondyloarthritis: 4-year results from the MEASURE 2, 3 and 4 phase III trials. Rheumatol Int. 2022 Feb;42(2):205-213. doi: 10.1007/s00296-021-05044-6. Epub 2021 Nov 13. PMID 34773130
- [Derived] van der Horst-Bruinsma I, Miceli-Richard C, Braun J, Marzo-Ortega H, Pavelka K, Kivitz AJ, Deodhar A, Bao W, Porter B, Pournara E. A Pooled Analysis Reporting the Efficacy and Safety of Secukinumab in Male and Female Patients with Ankylosing Spondylitis. Rheumatol Ther. 2021 Dec;8(4):1775-1787. doi: 10.1007/s40744-021-00380-2. Epub 2021 Oct 7. PMID 34618347
- [Derived] Schett G, Baraliakos X, Van den Bosch F, Deodhar A, Ostergaard M, Gupta AD, Mpofu S, Fox T, Winseck A, Porter B, Shete A, Gensler LS. Secukinumab Efficacy on Enthesitis in Patients With Ankylosing Spondylitis: Pooled Analysis of Four Pivotal Phase III Studies. J Rheumatol. 2021 Aug;48(8):1251-1258. doi: 10.3899/jrheum.201111. Epub 2021 Mar 15. PMID 33722947
- [Derived] Baraliakos X, Van den Bosch F, Machado PM, Gensler LS, Marzo-Ortega H, Sherif B, Quebe-Fehling E, Porter B, Gaillez C, Deodhar A. Achievement of Remission Endpoints with Secukinumab Over 3 Years in Active Ankylosing Spondylitis: Pooled Analysis of Two Phase 3 Studies. Rheumatol Ther. 2021 Mar;8(1):273-288. doi: 10.1007/s40744-020-00269-6. Epub 2020 Dec 22. PMID 33351179
- [Derived] Himmler S, Branner JC, Ostwald DA. The societal impact of a biologic treatment of ankylosing spondylitis: a case study based on secukinumab. J Comp Eff Res. 2021 Feb;10(2):143-155. doi: 10.2217/cer-2020-0077. Epub 2020 Nov 30. PMID 33252266
- [Derived] Kvien TK, Conaghan PG, Gossec L, Strand V, Ostergaard M, Poddubnyy D, Williams N, Porter B, Shete A, Gilloteau I, Deodhar A. Secukinumab and Sustained Reduction in Fatigue in Patients With Ankylosing Spondylitis: Long-Term Results of Two Phase III Randomized Controlled Trials. Arthritis Care Res (Hoboken). 2022 May;74(5):759-767. doi: 10.1002/acr.24517. Epub 2022 Mar 10. PMID 33227175
- [Derived] Deodhar AA, Miceli-Richard C, Baraliakos X, Marzo-Ortega H, Gladman DD, Blanco R, Das Gupta A, Martin R, Safi J Jr, Porter B, Shete A, Rosenbaum JT. Incidence of Uveitis in Secukinumab-treated Patients With Ankylosing Spondylitis: Pooled Data Analysis From Three Phase 3 Studies. ACR Open Rheumatol. 2020 May;2(5):294-299. doi: 10.1002/acr2.11139. Epub 2020 Apr 30. PMID 32352653
- [Derived] Deodhar A, Gladman DD, McInnes IB, Spindeldreher S, Martin R, Pricop L, Porter B, Safi J Jr, Shete A, Bruin G. Secukinumab Immunogenicity over 52 Weeks in Patients with Psoriatic Arthritis and Ankylosing Spondylitis. J Rheumatol. 2020 Apr;47(4):539-547. doi: 10.3899/jrheum.190116. Epub 2019 Jun 15. PMID 31203228
- [Derived] Braun J, Deodhar A, Landewe R, Baraliakos X, Miceli-Richard C, Sieper J, Quebe-Fehling E, Martin R, Porter B, Gandhi KK, van der Heijde D; MEASURE 1 and MEASURE 2 study groups. Impact of baseline C-reactive protein levels on the response to secukinumab in ankylosing spondylitis: 3-year pooled data from two phase III studies. RMD Open. 2018 Nov 21;4(2):e000749. doi: 10.1136/rmdopen-2018-000749. eCollection 2018. PMID 30564451
- [Derived] Wei JC, Baeten D, Sieper J, Deodhar A, Bhosekar V, Martin R, Porter B. Efficacy and safety of secukinumab in Asian patients with active ankylosing spondylitis: 52-week pooled results from two phase 3 studies. Int J Rheum Dis. 2017 May;20(5):589-596. doi: 10.1111/1756-185X.13094. Epub 2017 May 25. PMID 28544533
- [Derived] Marzo-Ortega H, Sieper J, Kivitz A, Blanco R, Cohen M, Martin R, Readie A, Richards HB, Porter B; Measure 2 Study Group. Secukinumab and Sustained Improvement in Signs and Symptoms of Patients With Active Ankylosing Spondylitis Through Two Years: Results From a Phase III Study. Arthritis Care Res (Hoboken). 2017 Jul;69(7):1020-1029. doi: 10.1002/acr.23233. Epub 2017 Jun 7. PMID 28235249
- [Derived] Sieper J, Deodhar A, Marzo-Ortega H, Aelion JA, Blanco R, Jui-Cheng T, Andersson M, Porter B, Richards HB; MEASURE 2 Study Group. Secukinumab efficacy in anti-TNF-naive and anti-TNF-experienced subjects with active ankylosing spondylitis: results from the MEASURE 2 Study. Ann Rheum Dis. 2017 Mar;76(3):571-592. doi: 10.1136/annrheumdis-2016-210023. Epub 2016 Aug 31. PMID 27582421
- [Derived] Baeten D, Sieper J, Braun J, Baraliakos X, Dougados M, Emery P, Deodhar A, Porter B, Martin R, Andersson M, Mpofu S, Richards HB; MEASURE 1 Study Group; MEASURE 2 Study Group. Secukinumab, an Interleukin-17A Inhibitor, in Ankylosing Spondylitis. N Engl J Med. 2015 Dec 24;373(26):2534-48. doi: 10.1056/NEJMoa1505066. PMID 26699169

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo subcutaneous injection once weekly at baseline, Weeks 1, 2, 3 and 4, followed by dosing every 4 weeks up to week 16
- Placebo - Secukinumab 75 mg: Placebo patients re-randomized to secukinumab 75 mg subcutaneous injection every 4 weeks starting from week 16.
- Placebo - Secukinumab 150 mg: Placebo patients re-randomized to secukinumab 150 mg subcutaneous injection every 4 weeks starting from week 16.
Period: Up to Week 16
Arm/Group | Secukinumab 75 mg | Secukinumab 150 mg | Placebo | Placebo - Secukinumab 75 mg | Placebo - Secukinumab 150 mg
Started | 73 | 72 | 74 | 0 | 0
Completed | 68 | 66 | 66 | 0 | 0
Not Completed | 5 | 6 | 8 | 0 | 0
Not completed — Adverse Event | 2 | 5 | 4 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Period: Week 16 up to Week 260
Arm/Group | Secukinumab 75 mg | Secukinumab 150 mg | Placebo | Placebo - Secukinumab 75 mg | Placebo - Secukinumab 150 mg
Started | 68 | 66 | 0 | 32 | 34
Completed | 48 | 53 | 0 | 20 | 29
Not Completed | 20 | 13 | 0 | 12 | 5
Not completed — Lack of Efficacy | 7 | 4 | 0 | 4 | 2
Not completed — Non-compliance | 0 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0
Not completed — Technical issues | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 2 | 0 | 3 | 1
Not completed — Death | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 2 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 75 mg | Secukinumab 150 mg | Placebo | Total
Number analyzed (Participants) | 73 | 72 | 74 | 219
Age, Customized [Number; unit: participants]
  < 65 years | 70 | 70 | 72 | 212
  >= 65 to 74 years | 2 | 2 | 1 | 5
  >= 75 years | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 18 | 66
  Male | 51 | 46 | 56 | 153
Race/Ethnicity, Customized [Number; unit: participants]
  White | 70 | 69 | 70 | 209
  Asian | 3 | 2 | 4 | 9
  American Indian or Alaska Native | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving ASAS 20 (SpondyloArthritis International Society Criteria) Response at Week 16
Description: ASAS 20 response is a validated composite assessment reflecting the percentage of treated patients who achieve within a defined timeframe an improvement of 20% and ≥1 unit on a scale of 1 to 10 in at least three of the four ASAS main domains and no worsening of ≥20% and ≥1 unit in the remaining domain. ASAS 20 is used to assess the efficacy of at least one dose of secukinumab against placebo.
Time Frame: Baseline up to 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab 75 mg | Secukinumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 72 | 74
percentage of participants | 41.1 | 61.1 | 28.4
Statistical Analysis 1: Comparison: Secukinumab 75 mg vs Placebo; Test type: Superiority; p = 0.0967, Regression, Logistic; Missing ASAS responses considered nonresponders; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.90 to 3.67]
Statistical Analysis 2: Comparison: Secukinumab 150 mg vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Missing ASAS responses considered nonresponders; Odds Ratio (OR) = 4.38, 95% CI 2-sided [2.14 to 8.96]

2. Secondary Outcome: Percentage of Participants Achieving ASAS 40 (SpondyloArthritis International Society Criteria) Response
Description: ASAS 40 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined timeframe an improvement of ≥40% and ≥2 units on a scale of 0 to 10 (0 being worse and 10 being better) in at least three of the four ASAS main domains (patient global, pain, function and inflammation) and no worsening at all in the remaining domain.
  ASAS 40 is used to assess the efficacy of at least one dose of secukinumab against placebo.
Time Frame: Baseline up to 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab 75 mg | Secukinumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 72 | 74
percentage of participants | 26.0 | 36.1 | 10.8
Statistical Analysis 1: Comparison: Secukinumab 75 mg vs Placebo; Test type: Superiority; p = 0.0194, Regression, Logistic; Missing ASAS responses considered nonresponders; Odds Ratio (OR) = 2.99, 95% CI 2-sided [1.19 to 7.48]
Statistical Analysis 2: Comparison: Secukinumab 150 mg vs Placebo; Test type: Superiority; p < .0004, Regression, Logistic; Missing ASAS responses considered nonresponders; Odds Ratio (OR) = 5.07, 95% CI 2-sided [2.06 to 12.44]

3. Secondary Outcome: Change From Baseline at Week 16 in Serum hsCRP
Description: The change from baseline in hsCRP is expressed as a ratio of post-baseline to baseline values. With the ratio normalized to 1.0 at baseline, ratios less than 1.0 represent decreased post-baseline values, whereas ratios greater than 1.0 represent increased post-baseline values. Blood levels of C-reactive protein (CRP), an acute phase reactant, are indicative of inflammation and of its severity, and can be used to monitor treatment response. A high sensitvity CRP (hsCRP) test is implemented in this study to assess the efficacy of at least one dose of secukinumab versus placebo in reducing AS elicited systemic inflammation over time.
Time Frame: Baseline up to 16 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Secukinumab 75 mg | Secukinumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 72 | 74
mg/L | 0.61 (1.103) | 0.55 (1.104) | 1.13 (1.105)
Statistical Analysis 1: Comparison: Secukinumab 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 0.54, 95% CI 2-sided [0.41 to 0.71]
Statistical Analysis 2: Comparison: Secukinumab 150 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 0.49, 95% CI 2-sided [0.37 to 0.64]

4. Secondary Outcome: Percentage of Participants Achieving ASAS 5/6 (SpondyloArthritis International Society Criteria) Response at Week 16
Description: ASAS 5/6 response is a validated composite assessment, reflecting the percentage of treated patients who achieve within a defined timeframe at least 20% improvement in score in at least 5 of a conventional set of 6 clinical domains relevant to AS (pain, patient global assessment, function, inflammation, spinal mobility, C-reative protein) without deterioration in the 6th domain. In this study, ASAS 5/6 is used to assess the efficacy of at least one dose of secukinumab against placebo.
Time Frame: Baseline up to 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab 75 mg | Secukinumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 72 | 74
percentage of participants | 34.2 | 43.1 | 8.1
Statistical Analysis 1: Comparison: Secukinumab 75 mg vs Placebo; Test type: Superiority; p = 0.0003, Regression, Logistic; Missing ASAS responses considered nonresponders; Odds Ratio (OR) = 6.13, 95% CI 2-sided [2.31 to 16.26]
Statistical Analysis 2: Comparison: Secukinumab 150 mg vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Missing ASAS responses considered nonresponders; Odds Ratio (OR) = 9.15, 95% CI 2-sided [3.47 to 24.12]

5. Secondary Outcome: Change From Baseline at Week 16 for Total Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: BASDAI is a validated assessment tool using 1 through 10 scales (1 indicating "no problem" and 10 indicating " worst problem"), to characterize six clinical domains (fatigue, spinal pain, joint pain/selling, localized tenderness, morning stiffness duration, morning stiffness severity) pertaining to five major symptoms of AS perceived by the patients. Computed composite scores of 4 or greater indicate suboptimal disease control. In this study, the BASDAI is used to assess the efficacy of at least one dose of secukinumab verus placebo.
Time Frame: Baseline up to 16 weeks
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 75 mg | Secukinumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 72 | 74
scores on a scale | -1.92 (0.249) | -2.19 (0.248) | -0.85 (0.252)
Statistical Analysis 1: Comparison: Secukinumab 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -1.07, 95% CI 2-sided [-1.77 to -0.37], Standard Error of Mean 0.353
Statistical Analysis 2: Comparison: Secukinumab 150 mg vs Placebo; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = -1.34, 95% CI 2-sided [-2.04 to -0.65], Standard Error of Mean 0.353

6. Secondary Outcome: Change From Baseline at Week 16 in Physical Function Component Summary (PCS) of the Medical Outcomes Study Questionnaire Short-form Health Survey (SF-36)
Description: Physical Function Component Summary (PCS) is only 1 component of SF-36. This scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Baseline up to 16 weeks
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 75 mg | Secukinumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 72 | 74
scores on a scale | 4.77 (0.798) | 6.06 (0.784) | 1.92 (0.786)
Statistical Analysis 1: Comparison: Secukinumab 75 mg vs Placebo; Test type: Superiority; p = 0.0110, Mixed Models Analysis; Mean Difference (Net) = 2.84, 95% CI 2-sided [0.66 to 5.03], Standard Error of Mean 1.108
Statistical Analysis 2: Comparison: Secukinumab 150 mg vs Placebo; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Mean Difference (Net) = 4.14, 95% CI 2-sided [1.96 to 6.32], Standard Error of Mean 1.105

7. Secondary Outcome: Change From Baseline at Week 16 in ASQoL
Description: ASQoL is an 18 item questionnaire that assesses disease-specific quality of life (QoL), consisting of statements that are relevant to the physical and mental conditions for a participant with AS: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each statement is answered by the participant as a 'Yes' (scored as 1) or 'No' (scored as 0). All item scores are summed to give a total score. Total score can range from 0 (good QoL) to 18 (poor QoL). In this study, ASQoL is used to assess improvement from baseline of at least one dose of secukinumab versus placebo.
Time Frame: Baseline up to 16 weeks
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 75 mg | Secukinumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 72 | 74
scores on a scale | -3.33 (0.537) | -4.00 (0.528) | -1.37 (0.530)
Statistical Analysis 1: Comparison: Secukinumab 75 mg vs Placebo; Test type: Superiority; p = 0.0096, Mixed Models Analysis; Mean Difference (Net) = -1.96, 95% CI 2-sided [-3.43 to -0.48], Standard Error of Mean 0.748
Statistical Analysis 2: Comparison: Secukinumab 150 mg vs Placebo; Test type: Superiority; p = 0.0005, Mixed Models Analysis; Mean Difference (Net) = -2.63, 95% CI 2-sided [-4.09 to -1.16], Standard Error of Mean 0.743

8. Secondary Outcome: Percentage of Participants Achieving ASAS Partial Remission at Week 16
Description: ASAS partial remission is a composite assessment, reflecting the proportion of treated patients who achieve within a defined time frame a value not above 2 units in each of the 4 ASAS domains on a scale 0 to 10. In this study ASAS partial remission is used to assess the efficacy of at least one dose of secukinumab versus placebo.
Time Frame: Baseline up to 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab 75 mg | Secukinumab 150 mg | Placebo
Number analyzed (Participants) | 73 | 72 | 74
percentage of participants | 15.1 | 13.9 | 4.1
Statistical Analysis 1: Comparison: Secukinumab 75 mg vs Placebo; Test type: Superiority; p = 0.0325, Regression, Logistic; Missing ASAS responses considered nonresponders; Odds Ratio (OR) = 4.28, 95% CI 2-sided [1.13 to 16.21]
Statistical Analysis 2: Comparison: Secukinumab 150 mg vs Placebo; Test type: Superiority; p = 0.0471, Regression, Logistic; Missing ASAS responses considered nonresponders; Odds Ratio (OR) = 3.91, 95% CI 2-sided [1.02 to 15.01]

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately up to 5.5 years
Groups:
- Any Secukinumab 75 mg: Includes patients originally randomized to secukinumab 75 mg at baseline and placebo patients who were re-randomized to secukinumab 75 mg at week 16 (AEs occurring after re-randomization).
- Any Secukinumab 150 mg: Includes patients originally randomized to secukinumab 150 mg at baseline, placebo patients re-randomized to secukinumab 150 mg at Week 16 (AEs occuring after re-randomization) and patients who up-titrated from secukinumab 75 mg to 150 mg (AEs occurring after up-titration).
- Placebo: Includes patients originally randomized to Placebo for AEs until the time of re-randomization (Week 16) to Secukinumab
Arm/Group | Any Secukinumab 75 mg | Any Secukinumab 150 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 2/105 | 1/155 | 0/74
Serious Adverse Events (participants affected / at risk) | 25/105 | 31/155 | 4/74
Other Adverse Events (participants affected / at risk) | 76/105 | 99/155 | 26/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any Secukinumab 75 mg (N=105) | Any Secukinumab 150 mg (N=155) | Placebo (N=74)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0
Iritis (Eye disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Drug ineffective (General disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0
Gallbladder abscess (Infections and infestations) | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Paraganglion neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 2 | 0
Quadriparesis (Nervous system disorders) | 0 | 1 | 0
Quadriplegia (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any Secukinumab 75 mg (N=105) | Any Secukinumab 150 mg (N=155) | Placebo (N=74)
Diarrhoea (Gastrointestinal disorders) | 9 | 17 | 1
Fatigue (General disorders) | 4 | 5 | 5
Bronchitis (Infections and infestations) | 15 | 14 | 1
Gastroenteritis (Infections and infestations) | 6 | 13 | 1
Influenza (Infections and infestations) | 13 | 14 | 0
Nasopharyngitis (Infections and infestations) | 30 | 35 | 3
Oral herpes (Infections and infestations) | 6 | 8 | 0
Pharyngitis (Infections and infestations) | 6 | 3 | 0
Rhinitis (Infections and infestations) | 6 | 5 | 1
Sinusitis (Infections and infestations) | 5 | 8 | 1
Upper respiratory tract infection (Infections and infestations) | 13 | 16 | 2
Urinary tract infection (Infections and infestations) | 5 | 9 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 | 8 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 6 | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 10 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 13 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 8 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 11 | 1
Dizziness (Nervous system disorders) | 2 | 3 | 4
Headache (Nervous system disorders) | 9 | 15 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 2
Rash (Skin and subcutaneous tissue disorders) | 6 | 4 | 1
Hypertension (Vascular disorders) | 9 | 15 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial